CLINICAL TRIAL: NCT00401011
Title: An Open-Label Phase I/II Study of the Safety and Efficacy of Perifosine and Bortezomib With or Without Dexamethasone for Patients With Relapsed or Refractory Multiple Myeloma Previously Treated With Bortezomib
Brief Title: Safety & Efficacy Study of Perifosine + Bortezomib +/- Dexamethasone for Multiple Myeloma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Perifosine 218
Record Dates: First submitted 2006-11-15; First posted 2006-11-17 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2012-02

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse
Keywords: Perifosine; Bortezomib; Dexamethasone; Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — perifosine; Bortezomib; Dexamethasone; Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: In the Phase I part, maximum tolerated dose (MTD) is determined in sequential cohorts of patients. All patients will start with perifosine and bortezomib (cf. arms and interventions). In case of progression, dexamethasone 20 mg will be added to treatment. Phase II: open-label single treatment arm.
Oversight: Data Monitoring Committee: No

ARMS (6):
- Phase II: Perifosine + Bortezomib (Experimental): All patients will start with perifosine at bedtime daily and Bortezomib IV on days 1, 4, 8, and 11 q 21 days. Patients will be evaluated at q 3 weeks. If the patient has a CR, PR, MR or stable disease, they will continue treatment.
  Interventions: Drug: Perifosine; Drug: Bortezomib
- Phase II: Perifosine + Bortezomib + Dexa (Experimental): If the patient shows progressive disease, dexamethasone 20 mg will be added on days 1, 2, 4, 5, 8, 9, 11, 12, 15, 16, 18, and 19 to perifosine at bedtime and bortezomib IV on days 1, 4, 8, and 11 q 21 days.
  Interventions: Drug: Perifosine; Drug: Bortezomib; Drug: Dexamethasone
- Phase I: Dose 1: Perifosine + Bortezomib (Experimental): Perifosine 50 mg at bedtime and bortezomib 1 mg/m2 on days 1, 4, 8, and 11 every 3 weeks.
  Interventions: Drug: Perifosine; Drug: Bortezomib
- Phase I: Dose 2: Perifosine + Bortezomib (Experimental): Perifosine 100 mg at bedtime and bortezomib 1 mg/m2 on days 1, 4, 8, and 11 every 3 weeks
  Interventions: Drug: Perifosine; Drug: Bortezomib
- Phase I: Dose 3: Perifosine + Bortezomib (Experimental): Perifosine 50 mg at bedtime and bortezomib 1.3 mg/m2 on days 1, 4, 8, and 11 every 3 weeks
  Interventions: Drug: Perifosine; Drug: Bortezomib
- Phase I: Dose 4: Perifosine + Bortezomib (Experimental): Perifosine 100 mg at bedtime and bortezomib 1.3 mg/m2 on days 1, 4, 8, and 11 every 3 weeks
  Interventions: Drug: Perifosine; Drug: Bortezomib

INTERVENTIONS:
Drug: Perifosine — Phase I: Patients will receive daily perifosine (doses 50 mg/m2 or 100 mg/m2) at bedtime.
  Phase II: All patients will receive daily perifosine at bedtime. Patients will be evaluated every 3 weeks.
  Other Names: D-21266; KRX-0401
Drug: Bortezomib — Phase I: Patients will receive 1 mg/m2 or 1.3 mg/m2 on days 1, 4, 8, and 11 every 3 weeks. Phase II: Patients will receive bortezomib on days 1,4,8 and 11 every 3 weeks.
  Other Names: Velcade
Drug: Dexamethasone — Phase II: If the patient shows progressive disease after 3 weeks, dexamethasone 20 mg will be added to perifosine and bortezomib on days 1, 2, 4, 5, 8, 9, 11, 12, 15, 16, 18, and 19 to perifosine at bedtime and bortezomib IV on days 1, 4, 8, and 11 q 21 days.
  Other Names: Dexa
  Arms: Phase II: Perifosine + Bortezomib + Dexa

SUMMARY:
This is a phase I/II study of perifosine in combination with bortezomib-with or without dexamethasone-for patients with relapsed or refractory multiple myeloma previously treated with bortezomib. The current protocol will enroll patients with relapsed or refractory multiple myeloma who have been previously treated with bortezomib. The patients will be treated with perifosine, 50 mg or 100 mg qhs, in combination with bortezomib to determine if there is any preliminary evidence that the addition of perifosine improves the outcome for these patients. Previous treatment with perifosine will be allowed in this study. Patients progressing on treatment with perifosine and bortezomib will receive dexamethasone 20 mg on days 1, 2, 4, 5, 8, 9, 11, 12, 15, 16, 18, and 19 of each 21-day cycle in addition to bortezomib and perifosine.

DETAILED DESCRIPTION:
The primary objective of the phase I portion is to determine the maximum tolerated dose of perifosine in combination with bortezomib in patients previously treated with bortezomib.

All patients will receive daily perifosine qhs with food. In the initial phase I study, 3 patients will be entered into a specified combination of perifosine and bortezomib cohorts. If no dose-limiting toxicity is observed, then three additional patients will be entered in cohort 4 - a full dose of bortezomib (1.3 mg/m2 on days 1, 4, 8 and 11 every 3 weeks). If this dose is tolerated it will be used for the phase II study, otherwise an intermediate dose of 1 mg/m2 on days 1, 4, 8, and 11 every 3 weeks will be employed.

The phase II study will use the maximum tolerated dose of bortezomib and perifosine. The primary objective of phase II portion is to determine the response rate (the combined CR + PR + MR) following treatment with perifosine + bortezomib in patients with multiple myeloma who have relapsed following initial front-line therapy, are refractory to their most recent therapy, and were previously treated with bortezomib. The secondary objectives of the phase II portion are;

1. To further assess the safety and tolerability of perifosine in combination with bortezomib-with or without dexamethasone-in patients with multiple myeloma.
2. To obtain correlative data in patients with multiple myeloma treated with perifosine in combination with bortezomib-with or without dexamethasone (NOTE Centers may choose not to participate in correlative studies).

ELIGIBILITY:
Inclusion Criteria:

1. Subject was previously diagnosed with multiple myeloma based on standard diagnostic criteria, as follows.

   Major criteria:
   * Plasmacytomas on tissue biopsy.
   * Bone marrow plasmacytosis (> 30% plasma cells).
   * Monoclonal immunoglobulin spike on serum electrophoresis immunoglobulin G (IgG) >3.5 g/dL or immunoglobulin A (IgA) > 2.0 g/dL; kappa or lambda light chain excretion > 1 g/day on 24 hour urine protein electrophoresis.

   Minor criteria:
   * Bone marrow plasmacytosis (10 to 30% plasma cells).
   * Monoclonal immunoglobulin present but of lesser magnitude than given under major criteria.
   * Lytic bone lesions.
   * Normal IgM < 50 mg/dL, IgA < 100 mg/dL or IgG < 600 mg/dL.
2. Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:
3. Any two of the major criteria.
4. Major criterion 1 plus minor criterion b, c, or d.
5. Major criterion 3 plus minor criterion a or c.
6. Minor criteria a, b, and c or a, b, and d.
7. Patients must have relapsed or refractory disease (refractory is defined as progression during treatment or within 60 days after the completion of treatment).
8. Patients must have been previously treated with bortezomib. Patients may have received prior perifosine.
9. Age >= 18 years at the time of signing informed consent document.
10. All necessary baseline studies for determining eligibility must be obtained within 14 days prior to enrollment. (Pregnancy test must be within 7 days for women of childbearing potential.)
11. Subject has an ECOG (Zubrod) performance status of 0 to 2.
12. Subject must be able to adhere to the study visit schedule and other protocol requirements.
13. Subject must understand and voluntarily sign an informed consent document.
14. Women of child-bearing potential (WCBP)- must have a negative serum or urine pregnancy test within 72 hours prior to enrollment. In addition, all sexually active WCBP and male patients must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study.

Exclusion Criteria:

1. Renal insufficiency (serum creatinine levels > 3 mg/dL).
2. Patients who present with either ALT or AST >= 2.5 X upper limit of normal (ULN) and/or patients with bilirubin >= 1.5 X ULN.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to perifosine (miltefosine or edelfosine).
4. Concomitant medications that include corticosteroids (except as indicated for other medical conditions or up to 100 mgs of hydrocortisone or equivalent as premedication for administration of certain medications or blood products), chemotherapy, or other therapy that is or may be active against myeloma within 2 weeks prior to Cycle 1 Day 1. Nitrosoureas must be discontinued 6 weeks prior to Cycle 1 Day 1.
5. Subjects with hemoglobin < 8.0 g/dL.
6. Subjects with an absolute neutrophil count (ANC) <= 500 cells/mm3.
7. Peripheral neuropathy of grade 3 or greater. Patients with painful grade 2 neuropathy are also excluded.
8. Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count >= 50,000 cells/mm3).
9. Previous history of intolerance of bortezomib or perifosine.
10. Any condition, including laboratory abnormalities, that in the opinion of the investigator places the subject at unacceptable risk if he/she were to participate in the study.
11. WCBP who are pregnant or breast-feeding or men and women who are not using adequate contraception.
12. Plasma cell leukemia at time of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose (MTD). Phase II: To determine response rate. | Every 3 weeks
  Phase I: To determine the MTD of perifosine in combination with bortezomib in patients previously treated with bortezomib.
  Phase II: The primary endpoint of the study was 6-month progression-free survival.

SECONDARY OUTCOMES:
Phase II: Tolerability and Safety | Every 3 weeks
  To assess the safety and tolerability of perifosine in combination with bortezomib - with or without dexamethasone.
Phase II: Correlative data | Every 3 weeks
  To obtain correlative data in patients with multiple myeloma treated with perifosine in combination with bortezomib-with or without dexamethasone

CONTACTS AND LOCATIONS:
Overall Officials: Paul Richardson, MD, Principal Investigator — Dana-Farber Cancer Institute

REFERENCES:
- [Result] Richardson PG, Wolf J, Jakubowiak A, Zonder J, Lonial S, Irwin D, Densmore J, Krishnan A, Raje N, Bar M, Martin T, Schlossman R, Ghobrial IM, Munshi N, Laubach J, Allerton J, Hideshima T, Colson K, Poradosu E, Gardner L, Sportelli P, Anderson KC. Perifosine plus bortezomib and dexamethasone in patients with relapsed/refractory multiple myeloma previously treated with bortezomib: results of a multicenter phase I/II trial. J Clin Oncol. 2011 Nov 10;29(32):4243-9. doi: 10.1200/JCO.2010.33.9788. Epub 2011 Oct 11. PMID 21990396